CLINICAL TRIAL: NCT07023367
Title: Parent Navigator Program (PNP) to Improve Outcomes in Latino/x Children and Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Nhu Tran, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHLA-25-00190
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Parent Navigator Program; Latino/x Children; High-Risk Infant Follow-up (HRIF); Early Intervention (EI); Neurodevelopmental Outcomes
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parent Navigator Program (Experimental)
  Interventions: Behavioral: Parent Navigator Program
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Parent Navigator Program — Participants in this group will be connected with a parent with lived experience to help get them obtain developmental follow up services and early intervention.
  Arms: Parent Navigator Program
Behavioral: Standard of Care — The families in the standard care group will have their connections to neurodevelopmental (ND) follow-up and support delivered in the standard fashion which consists of a referral to high-risk infant follow-up (HRIF) by discharge coordinator.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to see if a Parent Navigator Program (PNP) is helpful for Latino/x parents of babies with congenital heart disease (CHD) to get connected to developmental follow-up services. The main question it aims to answer are:

* Do families assigned to the Parent Navigator Program (PNP) have higher rates of connection to High-Risk Infant Follow-Up (HRIF)/Early Intervention (EI) compared to the standard care group 6 months after randomization?
* Do children assigned to the Parent Navigator Program (PNP) have better neurodevelopmental outcomes (NDOs) compared to the standard care group 6 months after randomization?
* Do parents assigned to the Parent Navigator Program (PNP) have decreased parental stress compared to the standard care group?

Researchers will compare the Parent Navigator group to the standard care group to see if parent navigator group is helpful in connecting families to High-Risk Infant Follow-Up (HRIF)/Early Intervention (EI), improving neurodevelopmental outcomes (NDOs), and lowering parental stress.

Participants will:

* Undergo developmental assessments and survey at newborn stage and at 6 months
* Participants randomly assigned to the Parent Navigator group will have weekly (at least) phone calls with the parent navigator
* Participants randomly assigned to the Parent Navigator group will complete a 30-minute phone interview about their experience with the parent navigator program 6 months after random assignment

ELIGIBILITY:
Latino/x Infants:

Inclusion Criteria:

* Infants born with CHD requiring medical/surgical intervention at less than 30 days of age
* Identify as Latino/x

Exclusion Criteria:

* Presence of a major genetic syndrome
* Intraventricular hemorrhage or other major structural brain lesion
* Undergoing end of life care

Parents of Latino/x Infants:

Inclusion Criteria:

* Identify as Latino/x

Exclusion Criteria:

* Not fluent in English or Spanish

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Total number of Visits to the High Risk Infant Follow Up clinic and Early Intervention between Parent Navigator Program and Standard of Care | Baseline to 6 months
  Each group's number of visits to the High Risk Infant Follow Up clinic will be counted using electronic medical record chart abstraction. Each group's number of Early Intervention visits will be counted using the Medical Abstraction Form, a self-report survey developed by the principal investigator that will be completed by parents. Parents will be asked how frequently they see the early interventionist and when the visits started, allowing for a calculation of the total number of visits.
Group comparison of neurodevelopmental outcomes measured by the Bayley Scales of Infant and Toddler Development | Baseline to 6 months
  Each infant in both arms of the study will be evaluated using the Bayley Scales of Infant and Toddler Development - 4th Edition at 6 months of age. Scores in cognitive, language, and motor domains will be obtained. Separate multiple linear regression analyses to examine group association with standard scores in each of the three domains (cognitive, language, and motor). Standard scores on the Bayley Scales of Infant and Toddler Development - 4th Edition are scaled to a metric with a mean of 100 and a standard deviation of 15. Standard scores range from 45 to 155, with 45 corresponding to a score below the 0.1st percentile and 155 corresponding to a score above the 99.9th percentile.
Average parental stress score over 6 months measured by the Parental Stress Scale | Baseline to 6 months
  Each parent in both arms of the study will complete the Parental Stress Scale at the two visits. Repeated measures analysis of variance or mixed model for repeated measures will be used to compare average parental stress between the groups over time. Scores on the Parental Stress Scale range from 18 to 90, with 18 indicating low stress and 90 indicating high stress.

CONTACTS AND LOCATIONS:
Overall Officials: Nhu Tran, PhD, RN, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No